CLINICAL TRIAL: NCT03030846
Title: Zahra Teymuri, Zahedan University of Medical Sciences
Brief Title: Investigation the Effects of Stabilization Exercises on Pain, Disability and Activity of Pelvic Floor Muscles in Patients With Postpartum Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Teymuri, zahra teymuri, Zahedan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZAUMS
Record Dates: First submitted 2017-01-15; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Postpartum Lumbopelvic Pain
Keywords: pregnancy; pelvic floor muscles; Lumbo-pelvic pain; Stabilization exercises; abdominal muscles thickness; Multifidus muscles thickness; Multifidus muscles cross section area
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- stabilization exercises (Experimental): stabilization exercises for 6 weeks, 3 sessions per week and each session was 40 minutes for the training group.
  Interventions: Other: Stabilization exercise
- control group (Experimental): electrotherapy include of 20 minutes TENS conventional and Ultrasound pulse for 10 minutes without any exercises for the control group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Stabilization exercise — 18 sessions during 6 consecutive weeks, three times per week, 30 or 40 minutes per session including: Twenty minutes for receiving hot pack and TENS and 10 or 20 minutes for training the exercises in 7 level : 1.Train the specific contraction of the deep abdominal muscles, multifidus and pelvic floor muscles(PFM). 2.Train the specific contraction of deep abdominal muscles with coactivation of multifidus and PFM in supine, prone, sitting, standing and quadruped position. 3. Segmental control exercises in close kinematic chain. 4. Segmental control exercises in open kinematic chain with limb loading, emphasis on abdominal muscles. 5. Segmental control exercises in open kinematic chain with limb loading, emphasis on back extensor muscles. 6. Progress exercises to functional task. 7. Coactivation of abdominal and multifidus muscles with limb loading in aerobic tasks.
  Arms: stabilization exercises
Other: Control group — 8 sessions during 6 consecutive weeks, three times per week, per session including: Twenty minutes for receiving hot pack and TENS
  Arms: control group

SUMMARY:
The purpose of this study was to evaluate the effects of stabilization exercises on pain, disability and pelvic floor muscles function in patients with lumbopelvic pain.

DETAILED DESCRIPTION:
Pregnancy is a specific experience that leads to several physical changes in women's body and influence most aspects of their lives. Pregnancy and delivery can cause serious complications such as urinary incontinence, pelvic organ prolapse, fecal incontinence, and low back pain (LBP) that have negative effects on women's sexual, physical, social and psychological health.

Based on Wu et al. systematic review, prevalence of pregnancy related low back pain (PLBP) during pregnancy and postpartum is 45% and 25% respectively.

LBP is one of the most current causes of disability and sick leave after delivery.Abnormal load transfer in the lumbopelvic region has been considered as one possible explanation to lumbopelvic pain.The local stabilizing muscles, i.e. the transversely oriented abdominal, diaphragm, the lumbar MF and the PFM Play an important role in load transfer in the lumbopelvic region.so, we considered that an exercise program that addresses muscular dysfunction, such as lumbar stabilization exercise can improve motor pattern of local stabilizing muscles and can use in management of postpartum lumbopelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old
* pain located between costal margin to gluteal fold with or without radiation to lower limbs
* onset of pain during pregnancy or after delivery
* history of delivery at least 3 months ago.

Exclusion Criteria:

* known chronic rheumatologic or Orthopedic disorders
* systemic locomotor disease
* history of fracture, neoplasm,intervertebral disk pathology or radiculopathy, spondylolysis or spondylolysthesis
* contraindication of exercises, heart disease, diabetes, thrombophlebitis, uncontrolled epilepsy
* ongoing pregnancy
* treatment with specific stabilisation exercise during previous 3 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
pain | 6 weeks
  Visual Analog Scale(VAS) questionnaire
Disability | 6 weeks
  Oswestry Disability Index(ODI) questionnaire
Pelvic Floor Muscle activity | 6 weeks
  Transabdominal approach of Ultrasound imaging
Abdominal muscles(Transverse Abdominis,Internal Oblique,External Oblique) thickness | 6 weeks
  Ultrasound imaging
Multifidus muscle thickness and crass section area(S1 level) | 6 weeks
  Ultrasound imaging

OTHER OUTCOMES:
age | 6 weeks
  with questionnaire
weight | 6 weeks
  with questionnaire
height | 6 weeks
  with questionnaire
Body Mass Index(BMI) | 6 weeks
  with questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Zahra Teymuri, Sistan and Bluchestan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teymuri Z, Hosseinifar M, Sirousi M. The Effect of Stabilization Exercises on Pain, Disability, and Pelvic Floor Muscle Function in Postpartum Lumbopelvic Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Dec;97(12):885-891. doi: 10.1097/PHM.0000000000000993. PMID 29979205